CLINICAL TRIAL: NCT02787850
Title: CoolSculpting the Abdomen Using an Applicator With a Crown Cooling Insert
Brief Title: CoolSculpting in the Abdomen Using Applicator With and Without CCI
Acronym: CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZA16-002
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-02

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CoolSculpting Treatment Cohort A (Experimental): Cohort A will be treated on one side of the abdomen (Abdominal side 1) at a protocol-defined temperature for 60 minutes using the CoolMax applicator without the Crown Cooling Insert. The contralateral side (Abdominal side 2) will be treated with the Crown Cooling Insert at a second protocol-defined temperature for 45 minutes.
  Each half of the abdominal area will be treated once, for a total of two treatments per subject.
  Interventions: Device: CoolSculpting Treatment
- CoolSculpting Treatment Cohort B (Active Comparator): Cohort B will be treated on one side of the abdomen (Abdominal side 1) at a protocol-defined temperature for 45 minutes using the CoolMax applicator with the Crown Cooling Insert. The contralateral side (Abdominal side 2) will be treated with a second protocol-defined temperature for 60 minutes with the Crown Cooling Insert.
  Each half of the abdominal area will be treated once, for a total of two treatments per subject.
  Interventions: Device: CoolSculpting Treatment

INTERVENTIONS:
Device: CoolSculpting Treatment — The CoolSculpting device will be used to perform treatments.

SUMMARY:
Evaluate the safety and efficacy of non-invasive subcutaneous fat layer reduction in the abdomen using an applicator with the Crown Cooling Insert.

DETAILED DESCRIPTION:
Evaluation of CoolSculpting treatment in the abdomen using a vacuum applicator with an accessory insert.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects >22 years of age and < 65 years of age.
* Subject has clearly visible fat on the abdomen, which in the investigator's opinion, may benefit from the treatment.
* Subject is a candidate for a standard CoolSculpting treatment with a CoolMax applicator.
* No weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed the study written informed consent form. Exclusion Criteria
* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system or any other metal containing implant.
* Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject has a history of hernia in the areas to be treated.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Subject is prone to severe claustrophobia (during MRI scans).
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leyda Bowes, MD, Principal Investigator — Bowes Dermatology Group
Locations (1):
- Bowes Dermatology Group, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects seeking reduction of fat in the abdomen were recruited from the general population.
Groups:
- CoolSculpting Treatment Cohort A: CoolSculpting device with and without Crown Cooling Insert and standard applicator and will be used to perform treatments on contralateral sides of the abdomen. Cohort A will receive treatments on one side of the abdomen without the Crown Cooling Insert with a protocol-defined temperature for 60 minutes. The contralateral side of the abdomen will be treated with the Crown Cooling Insert using a protocol-defined temperature for 45 minutes.
- CoolSculpting Treatment Cohort B: CoolSculpting device with the Crown Cooling Insert and standard applicator and will be used to perform treatments on contralateral sides of the abdomen. Cohort B subjects will be treated one one half of the abdomen with the Crown Cooling Insert at a protocol-defined temperature for 45 minutes. The contralateral side of the abdomen will also be treated with the Cron Cooling Insert at a protocol-defined temperature for 60 minutes.
Period: Overall Study
Arm/Group | CoolSculpting Treatment Cohort A | CoolSculpting Treatment Cohort B
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Contralateral sides of each subject's abdomen treatment using protocol-defined.temperatures and time. Cohort A will receive treatment on half of the abdomen using the Crown Cooling Insert; the contralateral half will be treated with the Crown Cooling Insert. Cohort B will be treated with the Crown Cooling Insert on both halves of the abdomen.
Groups:
- CoolSculpting Treatment Cohort A; CoolSculpting Treatment Cohort B: The treatments are designed to see if fat can be reduced in the abdomen with an applicator design incorporating a new insert. Treatment duration and cooling will vary between treatment sites and cohorts.
  The CoolSculpting device will be used to perform treatments.
- Total: Total of all reporting groups
Arm/Group | CoolSculpting Treatment Cohort A | CoolSculpting Treatment Cohort B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 44.4 [28 to 58] | 36.2 [22 to 53] | 40.3 [22 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Accurately Identified Pre-treatment Photos
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as at least 70% correct identification of pre-treatment images by two out of three reviewers.
Time Frame: 12 weeks post treatment
Population: The analysis population consisted of 19 subjects with evaluable images. Six images from each subject's abdomen were reviewed by the independent reviewers.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Groups:
- Overall Study Population-Both Cohorts: The analysis population included subjects enrolled in both cohorts of the study.
- Abdomen Site Treated Using CCI for 60 Minutes and Warmer Temperature: The abdomen was treated for a duration of 60 minutes per a protocol-defined temperature using the CCI applicator accessory.
- Abdomen Sites Treated With CCI for 45 Minutes: 1 side of the abdomen was treated for 45 minutes at a protocol defined temperature with the CCI applicator accessory.
- Abdomen Site Treated for 60 Minutes: One abdomen site was treated with a lower protocol-defined temperature for 60 minutes with the CCI accessory.
Arm/Group | Overall Study Population-Both Cohorts | Abdomen Site Treated Using CCI for 60 Minutes and Warmer Temperature | Abdomen Sites Treated With CCI for 45 Minutes | Abdomen Site Treated for 60 Minutes
Number analyzed (Participants) | 19 | 10 | 19 | 9
Number analyzed (photos) | 38 | 30 | 57 | 27
photos | 33 | 23 | 50 | 23
Statistical Analysis 1: Comparison: Overall Study Population-Both Cohorts; Test type: Other; sucess proportion = 86.8, 95% CI 2-sided [71.9 to 95.6]
Statistical Analysis 2: Comparison: Abdomen Site Treated Using CCI for 60 Minutes and Warmer Temperature; Test type: Other; success proportion = 76.7, 95% CI 2-sided [57.7 to 90.1]
Statistical Analysis 3: Comparison: Abdomen Sites Treated With CCI for 45 Minutes; Test type: Other; success proportion = 87.7, 95% CI 2-sided [76.3 to 94.9]
Statistical Analysis 4: Comparison: Abdomen Site Treated for 60 Minutes; Test type: Other; success proportion = 85.2, 95% CI 2-sided [66.3 to 95.8]

2. Primary Outcome: Participants With Unanticipated Adverse Device Effects (UADE)
Description: The number of unanticipated device effects will be tabulated to assess safety of the device and applicator accessory (Crown Cooling Insert). Adverse event data is collected from the time of enrollment through the 12 week follow-up visit.
Time Frame: Enrollment through 12 weeks post-treatment
Population: Subjects who received CoolSculpting treatment for reduction of subcutaneous fat in the abdomen were included in the analysis population. Of the 20 subjects enrolled and treated, one subject withdrew prior to study completion.
Measure: Number; unit: UADEs
Groups:
- Cohort A: One side of the abdomen was treated using the CoolMax applicator and the Crown Cooling Insert for 60 minutes at a protocol-defined temperature. The contralateral side of the abdomen was treated was treated using the CoolMax applicator and Crown Cooling Insert for 45 minutes at a protocol-defined temperature.
- Cohort B: One side of the abdomen was treated with the CoolMax applicator and Crown Cooling Insert for 45 minutes at a protocol-defined temperature; the contralateral side of the abdomen was treated with the CoolMax applicator and the Crown Cooling Insert for 60 minutes at a protocol-defined temperature.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 9
UADEs | 0 | 0

3. Secondary Outcome: Subject Satisfaction Questionnaire
Description: Subject satisfaction with the treatment experience data will also be collected via a written questionnaire at the 12-week follow up visits. This questionnaire will be composed of 5-point Likert scale questions, as well as free-text responses. Subjects will be asked to determine overall satisfaction with the treatment. The choices will be: 1) very satisfied; 2) somewhat satisfied; 3) neither satisfied nor unsatisfied; 4) somewhat unsatisfied; 5) very unsatisfied.
Time Frame: 12 weeks post-final treatment
Population: Groups include per-protocol subgroups for Cohort A and Cohort B. 20 subjects were assigned treatment parameters in Subgroup 2; one (1) subject withdrew from the study prior to completion.
Measure: Count of Participants; unit: Participants
Groups:
- Subgroup 1 Treatment Parameters: Abdomen areas treated with CoolSculpting without the Crown Cooling Inser for 60 minutes.
- Subgroup 2 Treatment Parameters: Abdomen areas treated with CoolSculpting with the Crown Cooling Insert for 45 minutes at a protocol defined temperature
- Subgroup 3 Treatment Parameters: Abdomen areas treated with CoolSculpting and the Crown Cooling insert for 60 minutes at a protocol-defined temperature
Arm/Group | Subgroup 1 Treatment Parameters | Subgroup 2 Treatment Parameters | Subgroup 3 Treatment Parameters
Number analyzed (Participants) | 10 | 19 | 9
Participants
  Very visible to visible fat reduction | 8 | 16 | 8
  Results expected or more than expected | 7 | 14 | 7
  Satisfied to very satisfied with procedure | 9 | 17 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through the 12-week final follow-up visit.
Description: Adverse events (AE) will be assessed continuously throughout the study. An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device.
Groups:
- Cohort A-Abdomen Side 1: Cohort A will be treated on one side of the abdomen (Abdominal side 1) at a protocol-defined temperature for 60 minutes without the Crown Cooling Insert.
- Cohort A-Abdomen Side 2: Abdomen side 2 will be treated using the CoolMax applicator and the Crown Cooling Insert for 45 minutes at a protocol-defined temperature.
- Cohort B-Abdomen Side 1: Cohort B will be treated on one side of the abdomen (Abdominal side 1) at a protocol-defined temperature for 45 minutes with the CoolMax Applicator and Crown Cooling Insert.
- Cohort B- Abdomen Side 2: Abdomen side 2 will be treated with the CoolMAx applicator at a second protocol-defined temperature for 60 minutes, with the Crown Cooling Insert.
Arm/Group | Cohort A-Abdomen Side 1 | Cohort A-Abdomen Side 2 | Cohort B-Abdomen Side 1 | Cohort B- Abdomen Side 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-Abdomen Side 1 (N=10) | Cohort A-Abdomen Side 2 (N=10) | Cohort B-Abdomen Side 1 (N=10) | Cohort B- Abdomen Side 2 (N=10)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No